CLINICAL TRIAL: NCT04288622
Title: A Randomised Controlled Trial Using Experience Sampling Method as a Way to Improve Depressive and Anxiety Symptoms in Women at Risk of Common Mental Disorder in Hong Kong
Brief Title: ESM-derived Personalised Feedback for Women at Risk of Common Mental Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yi-Nam Suen, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESM iCMD RCT
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Women at Risk of Common Mental Disorders
Keywords: Experience Sampling Method; At risk; Depression; Women; Randomized Controlled Trials; Feedback; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESM-derived personalised feedback (ESM-F) group (Experimental): Participants will be required to participate in an ESM data collection procedure. Participants will be required to complete a beep-questionnaire 3 days a week, over a 6-week period. The mobile app will be programmed to emit a beep 10 times per day at random intervals between 7.30 and 22.30. At each beep, participants will use the app to digitally complete a brief beep-questionnaire, which covers current affect, current context and activities. Moreover, participants will receive weekly standardized feedback on personalized patterns of positive affect.
  Interventions: Other: Weekly standardised, personalised feedback
- ESM group (No Intervention): Participant will be required to participate in the same ESM data collection procedure as the ESM-F group. The personalised feedback report will be given to the participant after the whole study period (32 weeks) instead of weekly during data collection process.
- Control (CON) group (No Intervention): Participants will not be required to participate in the 6-week ESM data collection procedure. They will also receive the personalised feedback report based on the ESM data collected at baseline and week 7.

INTERVENTIONS:
Other: Weekly standardised, personalised feedback — The ESM-F group will receive standardised ESM-derived feedback immediately followed the weekly ESM data collection procedure, totalling 6 times in the entire intervention period. The feedback will be provided by the researcher in the format of written report and verbal explanation. The feedback on participants' momentary affective state in specific daily life contexts and the association with depressive symptoms will be given. The changes in positive affect level and the number of depressive complaints over the course of the ESM intervention will be shown.
  Arms: ESM-derived personalised feedback (ESM-F) group

SUMMARY:
This study aims to examine the effectiveness of Experience Sampling Method (ESM) derived personalised feedback for women at risk of common mental disorder in Hong Kong, in reducing individuals depressive and anxiety symptoms.

DETAILED DESCRIPTION:
Women who are at-risk for common mental disorders and have completed the online screening for Jockey Club Mental Wellness Project for Women (JCWow) will be recruited. This study aims to test the effectiveness of ESM-derived personalized feedback in reducing symptoms of depression and anxiety using a randomised controlled trial. After given written consent, the participants will be required to undergo a 5 days baseline ESM data collection (week 0). Upon completion of baseline data collection, they will be randomly assigned to the intervention (ESM-F), active reference (ESM) or control (CON) group. The participants in the intervention group will participate in an ESM procedure (three days per week over a 6-week period) using through SMS system (week 1 - 6). This group will receive weekly standardised feedback on personalised patterns of positive affect. The active reference group will also participate in the same ESM procedure without a weekly feedback. The control group will not be required to undergo this 6-week data collection procedure. At week 7, all three groups will undergo another 5 days of post-intervention ESM data collection in order to examine the naturalistic and interventional changes on the depressive symptoms. From week 8 onwards, the participants will be contacted 5 times (week 8, 12, 16, 20 and 32) via telephone to follow-up their condition. After 32 weeks, both active reference and control group will receive the report.

ELIGIBILITY:
Inclusion Criteria:

* Women within the age range of 18-64
* Identified as at-risk for depressive disorders (iDD) using the Depression Subscale (scored 10 or above) in DASS-21
* Willing to provide written informed consent
* Understand Cantonese and can read or write Chinese
* Use a smartphone

Exclusion Criteria:

* Those mental conditions that require other treatment priorities (e.g., major depression, suicidal risk, substance abuse, current or past episodes of psychotic disorder, personality disorders).
* Those medical conditions that severely limit participation, comprehension, or adherence to treatment (e.g., epilepsy, dementia, terminal medical illness).
* Those who are receiving structured psychotherapy or counselling.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptoms | At week 32
  Measured by the Depression Subscale in Depression Anxiety Stress Scales (DASS-21). The subscale consists of 7 items, each with 4 options of responses (from 0-3), the total score of the subscale is calculated by summing up the item score of the 7 items and double it. It ranges from 0 to 42. Higher score indicates more severe level of depressive symptoms.
Severity of anxiety symptoms | At week 32
  Measured by the Anxiety Subscale in Depression Anxiety Stress Scales (DASS-21). The subscale consists of 7 items, each with 4 options of responses (from 0-3), the total score of the subscale is calculated by summing up the item score of the 7 items and double it. It ranges from 0 to 42. Higher score indicates more severe level of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Nam Suen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong